CLINICAL TRIAL: NCT05665790
Title: Study on Primary Lesion Treatment for Patients With Bone Metastases
Brief Title: Primary Lesion Treatment for Bone Metastases
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai 6th People's Hospital (Other)
Responsible Party: Principal Investigator, Zhao Hui, Principal Investigator, Shanghai 6th People's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20221202
Record Dates: First submitted 2022-12-18; First posted 2022-12-27 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Bone Metastases
MeSH Terms: interventions — Radiotherapy; Palliative Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- radiotherapy (Experimental)
  Interventions: Radiation: radiotherapy
- palliative surgery (Experimental)
  Interventions: Procedure: palliative surgery
- no primary leison treatment (No Intervention)

INTERVENTIONS:
Radiation: radiotherapy — radiotherapy
  Arms: radiotherapy
Procedure: palliative surgery — palliative surgery
  Arms: palliative surgery

SUMMARY:
This study will carry out a prospective cohort study to study the effect of different primary leison treatment modes on disease control, quality of life, economic cost and survival period of patients with bone metastases from breast cancer and lung cancer by giving radiotherapy or palliative surgery or not giving local treatment for the primary lesion in patients with bone metastases from breast cancer or lung cancer

ELIGIBILITY:
Inclusion Criteria:

1. HR positive breast cancer patients with bone metastasis or Non-small-cell lung cancer patients with bone metastasis；
2. Aged over 18;
3. ECOG：0-1；
4. Patients who benefit clinically(CR+PR) after 6 months of treatment.

Exclusion Criteria:

1. The expected life span is less than 3 months;
2. Have serious cardiovascular and cerebrovascular diseases, blood coagulation dysfunction, and cannot tolerate surgery;
3. Allergies to narcotic drugs;
4. The patient refused the treatment decision of the integrated team.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Disease control rate at 1 year | 1 year
  Disease control rate

SECONDARY OUTCOMES:
Progression-Free Survival | 1 year
Overall Survival | 1 year